CLINICAL TRIAL: NCT04474912
Title: Serum IL-17 Correlated With Inflammatory Changes But Not With Bony Changes in Both Hand Osteoarthritis and Rheumatoid Arthritis
Brief Title: Serum IL-17 Correlated With Inflammatory Changes in Osteoarthritis and Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Noha M Hammad, MD, Principal investigator, Zagazig University
Other Study IDs: 6293-22-7-2020
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis (RA) and Osteoarthritis (OA)
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Healthy volunteers with no symptoms or signs of rheumatoid arthritis or osteoarthritis
- Rheumatoid arthritis group: Rheumatoid arthritis (RA) patients fulfilled 2010 American college of rheumatology (ACR) classification criteria. A patient is considered having definite RA if he/she scores at least 6 points in the established classification system
- Osteoarthritis group: Osteoarthritis (OA) patients fulfilled 1990 ACR criteria for the classification and reporting of osteoarthritis of the hand. A patient is considered having hand OA if he /she Hand pain, aching, or stiffness plus 3 or 4 of hard tissue enlargement of 2 or more of 10 selected joints or hard tissue enlargement of 2 or more DIP joints or fewer than 3 swollen MCP joints, or deformity of at least 1 of 10 selected joints which are are the second and third distal interphalangeal (DIP), the second and third proximal interphalangeal, and the first carpometacarpal joints of both hands

SUMMARY:
The total number of the included subjects was 120 in 3 equal groups (RA, OA and control). All subject was subjected to serum IL17 level measurement. MSK US (of both wrists, MCPs, PIPs and DIPs) was done to all patients in RA and OA groups. Disease activity was measured by disease activity score (DAS28) for RA patients. Visual analogue scale for pain (VAS) was obtained from patients in RA and OA groups. Functional assessment was done using health assessment questionnaire (HAQ) for RA patients and the Australian/Canadian (AUSCAN) Osteoarthritis Hand Index for OA patients

ELIGIBILITY:
Inclusion Criteria:

* A patient is considered having definite RA if he/she scores at least 6 points in the established classification system
* A patient is considered having Hand OA if he /she Hand pain, aching, or stiffness plus 3 or 4 of hard tissue enlargement of 2 or more of 10 selected joints or hard tissue enlargement of 2 or more DIP joints or fewer than 3 swollen MCP joints, or deformity of at least 1 of 10 selected joints which are are the second and third distal interphalangeal (DIP), the second and third proximal interphalangeal, and the first carpometacarpal joints of both hands

Exclusion Criteria:

* Any subject with liver diseases, coronary artery diseases, kidney diseases or other inflammatory conditions was excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study participants will be recruited from attendants to Rheumatology and Rehabilitation outpatient clinic at Zagazig University Hospitals
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Clinical disease activity in Rheumatoid Arthritis (RA) and hand Osteoarthritis (OA) patients | 12 months
  During the whole course of the study, disease activity of the patients was measured by disease activity score (DAS28) for RA patients. Visual analogue scale for pain (VAS) was obtained from patients in RA and OA groups. Functional assessment was done using health assessment questionnaire (HAQ) for RA patients and the Australian/Canadian (AUSCAN) Osteoarthritis Hand Index for OA patients.

SECONDARY OUTCOMES:
IL-17 serum levels in RA and OA patients | 2 weeks
  IL-17 will be measured by enzyme linked immunosorbent assay from collected serum samples from the study participants

OTHER OUTCOMES:
Radiologic bony changes in RA and OA patients | 12 months
  During the whole course of the study period, recruited participants undergone musculoskeletal (MSK) ultrasound to assess the bony changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Faculty of Medicine, Zagazig, Sharqia Province, Egypt